CLINICAL TRIAL: NCT05153161
Title: Development of Memesto Wearable Repetitive Message/Music Therapy Device That Senses and Reduces Agitation in Alzheimer's Disease and Alzheimer's Disease Related Dementia (AD/ADRD) Individuals
Brief Title: Memesto Wearable Device for Persons With Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewater Safety Systems, Inc. (Industry)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R43AG074725-01 (NIH)
Record Dates: First submitted 2021-11-09; First posted 2021-12-10 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; ADRD; dementia; memory care; agitation; non-pharmacological intervention; medical device; SBIR; repetitive message therapy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Psychomotor Agitation

STUDY DESIGN:
Intervention Model Description: a proven protocol to test a pharmacological treatment of agitation in AD/ADRD persons using individuals in nursing homes and assisted care settings
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with ADRD living in a residential care facility (Experimental): Each consented participant will receive the current Memesto device and will be provided formal and informal training instructions. After consent and screening, a two-week training period with a Memesto device will be followed by ten weeks of data collection. An experienced research assistant will administer the baseline NPI in order to collect the agitation ratings by the family caregiver, and the professional caregiver will be collected by a trained research assistant and captured in an electronic case report form designed using REDCap.14,15 Then, participants will undergo evaluation of the NPI agitation domain at 2 weeks, 4 weeks, 6 weeks, 8 weeks, and 10 weeks. Adverse events related to the device will be collected from the family and professional caregivers. Human centered system designers will work with the operations team to enhance participant engagement and maintain high quality data collection.
  Interventions: Device: Memesto

INTERVENTIONS:
Device: Memesto — Edgewater plans to develop the next generation Memesto, a wearable device able to sense increasing agitation in ADRD sufferers and automatically deliver agitation-reducing personalized voice messages and music most effective at calming the individual based on past interventions. This innovative product will be the first wearable ADRD device to track agitation via body-worn sensors and automatically deploy agitation-reducing voice and music therapy without any caregiver interaction. The new system will use analytics to track the effectiveness of the various media and update the calming 'play list' over time.

SUMMARY:
An estimated 70% of the 7.2+ million people in the U.S. with Alzheimer's Disease and Alzheimer's Disease-Related Dementias experience agitation, characterized by poorly organized and purposeless psychomotor activity that diminishes their quality of life. The goal of this Small Business Innovation Research (SBIR) project is to develop a wearable therapy device that automatically senses rising agitation, and alerts caregivers while deploying calming voice and music therapy to help them avoid crisis level behavior. This device will improve health outcomes for AD/ADRD sufferers and reduce the substantial stress suffered by their caregivers.

DETAILED DESCRIPTION:
Edgewater Safety Systems developed a smart wearable media player (Memesto) that family and other caregivers could use with a web app to record, schedule and deliver voice and music to an ADRD patient through this device. Caregivers were able to record greetings, reminders to take medication, drink water or eat lunch, and these messages could be played for the patient via the device at set dates and times. In a follow-up survey with caregivers who used the Memesto with patients at care facilities, 11 of 11 rated it 4.5 out of 5 for "usefulness in mitigating agitation." Edgewater proposes to develop a more innovative wearable device that senses rising agitation in the patient and automatically plays therapeutic messages and music shown to have had the greatest success reducing or eliminating agitation in the wearer's previous episodes. With this next generation Memesto, Edgewater aims to improve quality of life for a diverse population of ADRD persons; diminish the use of potentially harmful drugs as an intervention; and help reduce stress and burnout in caregivers. The new Memesto will have four key elements of innovation: 1) repetitive, programmable voice and music therapy in a wearable device, a first for AD/ADRD care; 2) web-based app that enables family and friends to deliver personal messages and music anytime; 3) agitation-sensing system that reads biometric data from non-invasive body-worn sensors to automatically deploy media therapy; and 4) sensor data taken at start and end of the played media to determine effectiveness of that media in reducing agitation and continually prioritize the most effective media.In the Phase I study, Edgewater will partner with Rush Alzheimer's Disease Center to: 1) carry out a 10-week clinical trial on 20 ADRD persons to gather quantitative evidence of the original audio player's effectiveness at reducing agitation; and 2) demonstrate feasibility of ADRD agitation detection and automated intervention. Phase II will focus on complete implementation of a fully automated, miniaturized, wearable Memesto device and a broad field trial testing efficacy of the new agitation sensing and automated intervention system.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be adults with a dementia diagnosis who have clinically significant agitation, defined as a state of poorly organized and purposeless psychomotor activity characterized by at least one of the following: aggressive verbal (screaming, cursing), aggressive physical (destroying objects, grabbing, fighting), or non-aggressive physical (restlessness, pacing) behaviors.13 The behavioral symptoms must be severe enough to warrant pharmacological treatment. A family caregiver must be willing to participate along with a professional caregiver from the residential living facility.

Exclusion Criteria:

* Persons could screen fail if the device cannot be utilized by the person living with AD/ADRD, family caregiver, or professional caregiver.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 10 in average Neuropsychiatric Inventory (NPI) agitation domain score | 10 weeks
  The NPI agitation domain score is a composite score (symptom frequency x severity) ranging from 1 to 12; a higher score represents greater distress.

SECONDARY OUTCOMES:
Change from Baseline to Week 10 in average Clinical Global Impression - Severity (CGI-S) score | 10 weeks
  The CGI-S is rated on a 7-point Likert scale with responses ranging from 1 to 7; a higher score represents greater severity of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery T. Banker, MS, Principal Investigator — Edgewater Safety Systems, LLC
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Shah R, Basapur S, Hendrickson K, Anderson J, Plenge J, Troutman A, Ranjit E, Banker J. Does an Audio Wearable Lead to Agitation Reduction in Dementia: The Memesto AWARD Proof-of-Principle Clinical Research Study. Res Sq [Preprint]. 2025 Feb 17:rs.3.rs-6008628. doi: 10.21203/rs.3.rs-6008628/v1. PMID 40034447

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT05153161/Prot_SAP_000.pdf